CLINICAL TRIAL: NCT01452620
Title: Endovascular Abdominal Aortic Aneurysm Repair by Interventional Cardiologists
Acronym: EVAR
Status: Completed | Type: Observational
Sponsor: St. Joseph Mercy Oakland Hospital (Other)
Responsible Party: Principal Investigator, Abhijeet Basoor, MD, St. Joseph Mercy Oakland Hospital
Other Study IDs: 11-10-01
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Endovascular Abdominal Aortic Aneurysm Repair (EVAR)
Keywords: Endovascular Abdominal Aortic Aneurysm Repair (EVAR); Abdominal Aortic aneurysm (AAA)
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- EVAR cohort: All consecutive patients undergoing endovascular AAA repair (EVAR) in our community setting were followed for outcomes.

SUMMARY:
Registry for Endovascular repair of abdominal aortic aneurysm performed primarily by Interventional Cardiologists

ELIGIBILITY:
Inclusion Criteria:

* Patients with abdominal aortic aneurysm amenable for endovascular repair

Exclusion Criteria:

* Pregnant patients
* Patients less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study patients comprised of all patients undergoing endovascular abdominal aortic aneurysm repair performed primarily by Interventional Cardiologists in our community setting.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Mortality | mean follow up, 30 months

SECONDARY OUTCOMES:
Complications | mean follow up, 30 months
  Peri-procedural (30 day) and follow up complications

CONTACTS AND LOCATIONS:
Overall Officials: Abhijeet Basoor, MD, Principal Investigator — St. Joseph Mercy Oakland Hospital; Kiritkumar Patel, MD, Study Director — St. Joseph Mercy Oakland Hospital; Abdul R Halabi, MD, Study Director — St. Joseph Mercy Oakland Hospital; Nishit Choksi, MD, Study Director — St. Joseph Mercy Oakland Hospital; Thanh Phan, MD, Study Director — St. Joseph Mercy Oakland Hospital; Michele DeGregorio, MD, Study Director — St. Joseph Mercy Oakland Hospital
Locations (1):
- St. Joseph Mercy Oakland Hospital, Pontiac, Michigan, United States